CLINICAL TRIAL: NCT01334541
Title: A Brief Intervention to Reduce Suicide Risk in Military Service Members and Veterans- Study 1
Acronym: SAFE VET
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Columbia University (Other); University of Pennsylvania (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: W81XWH-09-2-0129-1
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2018-10

CONDITIONS: Suicide Risk | Patient

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SAFE VET
  Interventions: Behavioral: SAFE VET
- E-CARE

INTERVENTIONS:
Behavioral: SAFE VET — All SAFE VET EDs provide a standardized intervention that is specifically adapted for use in the ED to mitigate suicide risk. Given that the SAFE VET intervention was developed for use in a busy ED setting, the length of the intervention is approximately 45 minutes. The SAFE VET intervention is administered by a clinical provider who has been specifically trained and consists of:
  1. Risk Assessment
  2. Safety Planning Intervention: Developed by Stanley and Brown (2008), Safety Planning Intervention consists of a hierarchically-arranged list of coping strategies identified for use during a subsequent suicidal crisis.
  3. Clinical Follow-Up Protocol
  Groups: SAFE VET

SUMMARY:
The investigators propose to evaluate Suicide Assessment and Follow-up Engagement: Veteran Emergency Treatment (SAFE VET) which is currently being implemented in 4 VA ED/Urgent Care Units across the United States (Portland VA Medical Center (VAMC), Denver VAMC, Manhattan VAMC, and Philadelphia VAMC).

DETAILED DESCRIPTION:
Background: In 2009, a novel clinical demonstration project entitled Suicide Assessment and Follow-up Engagement: Veteran Emergency Treatment (SAFE VET) was initiated as a potential standard of care for suicidal Veterans who receive treatment at Veterans Affairs (VA) emergency departments (ED). SAFE VET is designed to attenuate suicide risk by helping Veterans manage suicidal thoughts and behaviors, and adhere to prescribed clinical care; thereby promoting resiliency and increased capacity to cope with suicidal states.

Objectives: Using a quasi-experimental design, the aim of this study is to compare the effectiveness of the SAFE VET intervention versus enhanced usual care (E-CARE)on the following: 1) the proportion of patients who attempt suicide within 6 months of index emergency department (ED) visit; 2) the severity of suicide ideation within 6 months after index ED visit; 3) the proportion of patients who attend > 1 outpatient mental health or substance abuse treatment appointments within 30 days following index ED visit; and 4) the degree of suicide-related coping for attending treatment during the 6 month period.

Methodology: Six hundred Veterans, up to 300 per condition (SAFE VET or E-CARE), who meet inclusion/exclusion criteria will be enrolled. E-CARE sites are as follows: Long Beach VAMC, Bronx VAMC, Milwaukee VAMC, and San Diego VAMC. All subjects will participate in an approximately 1-hour long baseline assessment battery (index ED visit) by phone, and will be contacted by phone at approximately 1, 3, and 6 months after the index ED visit to complete follow-up measures. Medical records will also be reviewed to determine VA health service usage in the six-month period after study enrollment.

ELIGIBILITY:
Inclusion Criteria:

Veterans will be enrolled who:

1. have received the SAFE VET intervention in VA SAFE VET EDs or treatment-as-usual in E-CARE EDs;
2. aged 18 years or older;
3. identified as being at risk for suicide based upon presenting complaints and/or the assessment of an ED clinician;
4. able to provide 2 contacts with telephone numbers for tracking purposes; and
5. able to provide a home/residential/shelter address where the participant resides and either a home, cellular, or other telephone number where the participant can be reached.

Exclusion Criteria:

Veterans will not be enrolled if they are:

1. unable to read and understand English;
2. unable or unwilling to give informed consent as determined either by the referring VA ED clinical staff or research personnel (see Mini Quiz below); and/or
3. admitted to the VA inpatient psychiatric unit from the ED.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who were seen in a VA Emergency Department and were identified as being at risk for suicide.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Columbia Suicide-Severity Rating Scale (C-SSRS; Posner et al., 2006; Posner et al. 2008). | Baseline and 1, 3, and 6 month follow-up assessments

SECONDARY OUTCOMES:
Scale for Suicide Ideation (SSI; Beck, Kovacs, & Weissman, 1979). | Baseline and 1, 3, and 6 month follow-up assessments

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Holloway, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences; Gregory Brown, Ph.D., Principal Investigator — University of Pennsylvania; Lisa Brenner, Ph.D., Principal Investigator — Denver VAMC, VISN 19 MIRECC; Barbara Stanley, Ph.D., Principal Investigator — Columbia University; Kerry Knox, Ph.D., Principal Investigator — Canadaigua VAMC- Center of Excellence; Glenn Currier, M.D., Principal Investigator — Canandaigua VAMC- Center of Excellence
Locations (8):
- United States (8):
  - Long Beach VAMC, Long Beach, California
  - San Diego VAMC, San Diego, California
  - Denver VAMC, Denver, Colorado
  - Manhattan VAMC, Manhattan, New York
  - Bronx VAMC, The Bronx, New York
  - Portland VAMC, Portland, Oregon
  - Philadelphia VAMC, Philadelphia, Pennsylvania
  - Milwaukee VAMC, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Matarazzo BB, Brown GK, Stanley B, Forster JE, Billera M, Currier GW, Ghahramanlou-Holloway M, Brenner LA. Predictive Validity of the Columbia-Suicide Severity Rating Scale among a Cohort of At-risk Veterans. Suicide Life Threat Behav. 2019 Oct;49(5):1255-1265. doi: 10.1111/sltb.12515. Epub 2018 Oct 9. PMID 30368871